CLINICAL TRIAL: NCT02161562
Title: OPTIMA: Efficacy of Optimized Re-treatment and Step-up Therapy With Omalizumab in CSU Patients
Brief Title: OPTIMA: Efficacy of Optimized Re-treatment and Step-up Therapy With Omalizumab in Chronic Spontaneous Urticaria (CSU) Patients
Acronym: OPTIMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIGE025ECA01
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: chronic spontaneous urticaria, CSU, chronic idiopathic urticaria, CIU, hives, angioedema, itch
MeSH Terms: conditions — Chronic Urticaria; Urticaria; Angioedema; Pruritus | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- omalizumab 150mg (Experimental): Participants received 150mg omalizumab every 4 weeks during the initial dosing phase (24 weeks). A second dosing period (at 150mg or 300mg) may have been implemented based on protocol-defined assessment criteria.
  Interventions: Drug: omalizumab
- omalizumab 300mg (Experimental): Participants received 300mg omalizumab every 4 weeks during the initial dosing phase (24 weeks). A second dosing period may have been implemented based on protocol-defined assessment criteria.
  Interventions: Drug: omalizumab

INTERVENTIONS:
Drug: omalizumab — 150mg omalizumab via sub-cutaneous injection once every 4 weeks
  Arms: omalizumab 150mg
Drug: omalizumab — 300mg omalizumab via sub-cutaneous injection once every 4 weeks
  Arms: omalizumab 300mg

SUMMARY:
This trial assessed the efficacy of optimized re-treatment therapy with omalizumab (150mg or 300mg) after relapse, in participants with Chronic Spontaneous Urticaria who were clinically well-controlled following their first course of treatment with omalizumab (150mg or 300mg). The study also assessed the benefit of uptitrating to 300mg dose in participants who were not well-controlled following their initial course of treatment with omalizumab 150mg, as well as the benefit of treatment extension of those patients who were not well-controlled following their initial course of treatment with omalizumab 300mg.

DETAILED DESCRIPTION:
The study consisted of 5 phases.

Phase 1 (Screening): At the first visit (Screening Visit), the participant was provided informed consent and then completed all screening visit assessments. During this visit, all CIU/CSU treatments taken by the participant were documented. Any protocol-defined prohibited CIU/CSU treatments were stopped at this visit, and the participant underwent a wash-out period of 1-5weeks (refer to study protocol for medication wash-out times) prior to Phase 2 Visit1. Only non-sedating H1- antihistamines, at locally-approved dosages, were allowed to be continued during the Screening Period and throughout the rest of the study. All participants also needed to complete daily diary during the entire screening period.

Phase 2 (Initial Dosing Period): Following completion of Phase 1, eligible participants were randomly assigned (in a 4:3 ratio) to either Group A or Group B. Participants in Group A were treated with omalizumab 150mg by subcutaneous (SC) injection every 4 weeks during the 24-week Phase 2 (Initial Dosing Period), while participants in Group B were treated with omalizumab 300mg every 4 weeks during this period. Randomization to treatment groups was stratified at Phase 2 Visit 1 by geographic location of the study site (i.e. Canada or Latin America), baseline presence/absence of angioedema and baseline UAS7 score (collected at Phase 2 Visit 1). At the end of Phase 2, all participants with a UAS7 score ≤ 6 entered Phase 3 (Study Treatment Withdrawal Period). Group A participants who had a UAS7 > 6 at any visit of Phase 2 starting at Week 8 (Phase2-Visit3) skipped Phase 3 and moved directly to Phase 4 (Second Dosing Period) and received 300 mg Omalizumab (step-up). Group B participants who had a UAS7 >6 at the end of Phase 2 skipped Phase 3 and moved directly to Phase 4.

Phase 3 (Study Treatment Withdrawal Period): During Phase 3 (Study Treatment Withdrawal Period), no study treatment (omalizumab) was given and participants continued to visit the study center at 4-week intervals (to a maximum of 8 weeks). If a UAS7 score ≥16 was observed during Phase 3 (Study Treatment Withdrawal Period), the participant moved directly to Phase 4 (Second Dosing Period). If a participant completed the full 8 weeks of Phase 3 (Study Treatment Withdrawal Period) with a UAS7 score <16, the participant was moved directly to Phase 5 (Follow-up Period).

Phase 4 (Second Dosing Period)

* Group A participants who relapsed (UAS7 ≥16) during Phase 3 (Study Treatment Withdrawal Period) were retreated with omalizumab 150mg by SC injection every 4 weeks during the 12-week Phase 4 (Second Dosing Period)
* Group A participants who were not clinically well-controlled at week 8 of Phase 2 (Initial Treatment Period) or any subsequent visit in Phase 2 moved to Phase 4 (Second Dosing Period) immediately during which their study treatment was up-titrated to 300mg by SC injection every 4 weeks for 12 weeks.
* Group A participants who had their symptoms well controlled at week 24 (UAS7≤6) but did not relapse during the 8 weeks Study Treatment withdrawal period (UAS7<16) moved directly to Phase 5, Follow up period.
* Group B participants who relapsed during Phase 3 (Study Treatment Withdrawal Period) were retreated with omalizumab 300mg by SC injection every 4 weeks during the 12- week Phase 4 (Second Dosing Period)
* Group B participants who were not clinically well-controlled at week 24 of Phase 2 (Initial Treatment Period) moved to Phase 4 (Second Dosing Period) immediately during which their study treatment remained 300mg by SC injection every 4 weeks for 12 weeks. In case the treating physician and the participant decided not to extend treatment, they could move directly from Phase 2 (Initial Treatment Period) to Phase 5 (Follow- up Period).
* Group B participants who had their symptoms well controlled at week 24 (UAS7≤6) but did not relapse during the 8 weeks Study Treatment withdrawal period (UAS7<16) moved directly to Phase 5, Follow up period.

Phase 5 (Follow-up Period)

* Participants who did not relapse (UAS7 <16) following completion of Phase 3 (Study Treatment Withdrawal Period) entered the 4-week Phase 5 (Follow-up Period).
* Group B participants who did not respond during their initial 24-week treatment period (Phase 2), and who did not wish to extend their treatment into Phase 4 (Second Dosing Phase) were allowed to move directly into the 4-week Phase 5 (Follow-up Period).
* All participants who completed Phase 4 (Second Dosing Period) entered the 4-week Phase 5 (Follow-up Period).

During Phase 5 (Follow-up Period), participants continued to only receive non-sedating H1- antihistamines at approved dosages. Omalizumab was not allowed to be administered during this period.

ELIGIBILITY:
Key Inclusion Criteria:

* Men or women at least 18 years of age at time of screening.
* Having a diagnosis of CSU and the presence of symptoms for ≥6 months prior to the screening visit.
* Presence of itch and hives for ≥6 consecutive weeks at any time prior to the screening visit despite concurrent use of non-sedating H1-antihistamine treatment
* Patient must have been on an approved dose of non-sedating H1-antihistamine for CSU, and no other concomitant CSU treatment, for at least the 7 consecutive days immediately prior to the randomization visit and must document current use on the day of the randomization visit.

Key Exclusion Criteria:

* Patients having a clearly defined underlying etiology for chronic urticaria other than CSU including the following urticarias: acute, solar, cholinergic, heat, cold, aquagenic, delayed pressure or contact
* Patients with other skin disease associated with itch that could interfere with study outcomes and/or compromise the safety of the patient
* Patients with evidence of parasitic infection
* Patients with a history of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Pregnant or nursing (lactating) women,
* Women of child-bearing potential, unless they are using effective methods of contraception during dosing of study treatment.
* Patients who are unable or unwilling to comply with study procedures, attend scheduled study visits, complete questionnaires and daily diaries, or who may otherwise be unable to comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-11-03 (Actual); Study Completion 2016-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- Argentina (5):
  - Novartis Investigative Site, Pilar, Buenos Aires
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Salta
- Brazil (4):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Alphaville / Barueri, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
- Canada (15):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, Markham, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Peterborough, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Toronto
- Novartis Investigative Site, Santiago, Chile
- Novartis Investigative Site, Santo Domingo, Republica Dominicana, Dominican Republic
- Novartis Investigative Site, Guatemala City, Guatemala
- Mexico (2):
  - Novartis Investigative Site, Zapopan, Jalisco
  - Novartis Investigative Site, Tlalpan, Mexico City
- Novartis Investigative Site, Panama City, Panama

REFERENCES:
- [Derived] Sussman G, Hebert J, Gulliver W, Lynde C, Yang WH, Papp K, Gooderham M, Chambenoit O, Khalil S, DeTakacsy F, Vieira A, Rihakova L. Omalizumab Re-Treatment and Step-Up in Patients with Chronic Spontaneous Urticaria: OPTIMA Trial. J Allergy Clin Immunol Pract. 2020 Jul-Aug;8(7):2372-2378.e5. doi: 10.1016/j.jaip.2020.03.022. Epub 2020 Apr 6. PMID 32272284

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomly assigned in a 4:3 ratio to Group A or Group B.
Groups:
- Omalizumab 150mg (A): Participants received 150mg omalizumab every 4 weeks during the initial dosing phase (24 weeks). A second dosing period (at 150mg or 300mg) may have been implemented based on protocol-defined assessment criteria.
- Omalizumab 300mg (B): Participants received 300mg omalizumab every 4 weeks during the initial dosing phase (24 weeks). A second dosing period may have been implemented based on protocol-defined assessment criteria.
Period: Overall Study
Arm/Group | Omalizumab 150mg (A) | Omalizumab 300mg (B)
Started | 178 | 136
Completed | 152 | 119
Not Completed | 26 | 17
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Protocol Violation | 9 | 4
Not completed — Pregnancy | 1 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Lack of Efficacy | 4 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Participant moved back to home country | 1 | 0
Not completed — Withdrew due to being out of the country | 1 | 0
Not completed — Participant moved out of province | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab 150mg (A) | Omalizumab 300mg (B) | Total
Number analyzed (Participants) | 178 | 136 | 314
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.7 (14.03) | 45.8 (13.60) | 46.3 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 99 | 229
  Male | 48 | 37 | 85

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Clinically Well-controlled (UAS7<=6) After the Initial Dosing Period, Relapsed (UAS7>=16) When Treatment Was Discontinued, and Who Achieved a UAS7 Score <=6 at the End of the Second Dosing Period (Retreatment A2 and B2)
Description: The UAS7 is a 7-day composite self-reported evaluation of itch (daily score 0-3) plus number of hives (daily score 0-3). The worst possible daily UAS score is 6, and the worst possible UAS7 score is 42. For this outcome, the participant's self-reported UAS7 score will be drawn from the last 7 days of the second dosing period.
Time Frame: Last 7 days of second dosing period, 44 weeks
Population: Participants from groups A2 (n=12) and B2 (n=44) were considered for the analysis. Only Groups A2 and B2 participants, who had UAS7 scores collected at end of the second dosing period, were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- All Retreatment (A2&B2): omalizumab 150 mg retreatment group + omalizummab 300 mg retreatment group
- Retreatment (A2): omalizumab 150 mg retreatment group
- Retreatment (B2): omalizumab 300 mg retreatment
Arm/Group | All Retreatment (A2&B2) | Retreatment (A2) | Retreatment (B2)
Number analyzed (Participants) | 49 | 12 | 37
Participants | 43 | 10 | 33

2. Secondary Outcome: The Difference in Urticaria Activity Score Over 7 Days (UAS7) Between the Start and End of the Second Dosing Period, in Participants That Step-up Treatment Dose During the Initial Dosing Period (Step-up A3)
Description: The UAS7 is a 7-day composite self-reported evaluation of itch (daily score 0-3) plus number of hives (daily score 0-3). The worst possible daily UAS score is 6, and the worst possible UAS7 score is 42. For this outcome, the participant's self-reported UAS7 score will be drawn from the 7 days prior to the second dosing period, and the last 7 days of the second dosing period. A negative change indicates improvement.
Time Frame: 7 days prior to start of second dosing period and last 7 days of Second Dosing Period
Population: Group A3 participants (n=141) were considered for the analysis. Only Group A3 participants, who had UAS7 scores collected at the start and end of the second dosing period, were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Step-up Treatment Group (A3): Step-up treatment from omalizumab 150 mg to 300 mg
Arm/Group | Step-up Treatment Group (A3)
Number analyzed (Participants) | 130
score on a scale | -9.5 (10.54)

3. Secondary Outcome: Number of Participants With Urticaria Activity Score Over 7 Days (UAS7)≤6 at the End of the Second Dosing Period, in Participants Who Stepped-up Treatment Dosing (Step-up A3)
Description: as for outcome 1
Time Frame: Last 7 days of the second dosing period
Population: Group A3 participants (n=141) were considered for the analysis. Only Group A3 participants, who had UAS7 scores collected at the end of the second dosing period, were analyzed.
Measure: Number; unit: Participants
Arm/Group | Step-up Treatment Group (A3)
Number analyzed (Participants) | 130
Participants | 59

4. Secondary Outcome: Time to Relapse (Urticaria Activity Score Over 7 Days (UAS7) ≥ 16) After Drug Withdrawal in Participants Who Responded to Initial Dosing Period (Retreatment A2 and B2)
Description: The UAS7 is a 7-day composite self-reported evaluation of itch (daily score 0-3) plus number of hives (daily score 0-3). The worst possible daily UAS score is 6, and the worst possible UAS7 score is 42. For this outcome, the time between end of initial dosing period to first occurence of UAS7 ≥ 16 will be evaluated.
Time Frame: study drug withdrawal period, weeks 24 through 32
Population: The Retreatment participants were analyzed (A2=12, B2=44).
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | All Retreatment (A2&B2) | Retreatment (A2) | Retreatment (B2)
Number analyzed (Participants) | 56 | 12 | 44
Weeks | 4.7 (2.37) | 4.8 (2.70) | 4.7 (2.31)

5. Secondary Outcome: Difference in Urticaria Activity Score Over 7 Days (UAS7) Between End of Initial Dosing Period and the End of the Second Dosing Period, in Group B3 Participants Who Did Not Respond to the Initial Dosing Period
Description: The UAS7 is a 7-day composite self-reported evaluation of itch (daily score 0-3) plus number of hives (daily score 0-3). The worst possible daily UAS score is 6, and the worst possible UAS7 score is 42. For this outcome, the participant's self-reported UAS7 score will be drawn from the last 7 days of the initial dosing period and the last 7 days of the second dosing period. A negative change indicates improvement.
Time Frame: last 7 days of initial dosing period, week 24, and last 7 days of second dosing period, week 36
Population: Group B3 participants (n=43) were considered for the analysis. Only B3 participants, who had UAS7 scores collected at both weeks 24 and 44, were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Extended Treatment (B3): omalizumab 300 mg extended treatment
Arm/Group | Extended Treatment (B3)
Number analyzed (Participants) | 41
score on a scale | -2.0 (10.50)

6. Secondary Outcome: The Change in Urticaria Activity Score Over 7 Days (UAS7) From Baseline to Week 24 in Group B Participants
Description: The UAS7 is a 7-day composite self-reported evaluation of itch (daily score 0-3) plus number of hives (daily score 0-3). The worst possible daily UAS score is 6, and the worst possible UAS7 score is 42. For this outcome, the participant's self-reported UAS7 score will be drawn from the 7-day period prior to Baseline visit and the last 7 days prior to the week 24 visit of initial dosing period. A negative change from baseline indicates improvement.
Time Frame: 7 days prior to Baseline visit, and last 7 days prior to week 24 of the initial dosing period
Population: Group B participants (n=136) were considered for the analysis. Only Group B participants, who had both baseline and week 24 UAS7 scores collected, were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omalizumab 300mg (B)
Number analyzed (Participants) | 131
score on a scale | -23.8 (10.08)

7. Secondary Outcome: Change in Urticaria Activity Score Over 7 Days (UAS7) Between Baseline and End of Second Dosing Period
Description: The UAS7 is a 7-day composite self-reported evaluation of itch (daily score 0-3) plus number of hives (daily score 0-3). The worst possible daily UAS score is 6, and the worst possible UAS7 score is 42. For this outcome, the participant's self-reported UAS7 score will be drawn from the 7 days before Baseline and the last 7 days of the second dosing period.
Time Frame: 7 days prior to Baseline visit, and last 7 days of second dosing period
Population: Group A (n=178) and Group B (n=136) participants were considered for the analysis. Only Group A and Group B participants who had both baseline and week 44 UAS7 scores collected, were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omalizumab 150mg (A) | Omalizumab 300mg (B) | Overall (A&B)
Number analyzed (Participants) | 156 | 122 | 278
score on a scale | -18.7 (11.66) | -23.0 (10.92) | -20.6 (11.53)

8. Secondary Outcome: The Number of Participants Who Remained Well-controlled (UAS7<=6) or Who Had Achieved UAS=0 at Phase 4 (Second Dosing Period) Week 8 During Retreatment After Being Well Controlled or Achieving UAS7=0 at Phase 2 (Initial Dosing Period) Week 8
Description: The UAS7 is a 7-day composite self-reported evaluation of itch (daily score 0-3) plus number of hives (daily score 0-3). The worst possible daily UAS score is 6, and the worst possible UAS7 score is 42. For this outcome, the participant's self-reported UAS7 score will be drawn from week 8 of initial dosing phase and week 8 of second dosing phase.
Time Frame: Week 8 of initial dosing phase and week 8 of second dosing phase
Population: Only Groups A2 and B2 participants, who had UAS7 scores collected at week 8 of initial dosing period and week 8 of second dosing period, were analyzed.
Measure: Number; unit: Participants
Arm/Group | All Retreatment (A2&B2) | Retreatment (A2) | Retreatment (B2)
Number analyzed (Participants) | 56 | 12 | 44
Participants
  UAS7<=6 at week 8 of the initial dosing period | 43 | 12 | 31
  UAS7=0 at week 8 of the initial dosing period | 34 | 10 | 24
  UAS7<=6 at week 8 of the second dosing period | 36 | 9 | 27
  UAS7=0 at week 8 of the second dosing period | 23 | 5 | 18

ADVERSE EVENTS:
Description: The serious adverse events (SAEs) count for the overall B group = 8 but the sum of the subgroups = 7. Per protocol, the subgroup assignment is based on the UAS7 outcome. The discrepancy mentioned previously is due to the fact that one participant was not assigned to a B subgroup because this participant was discontinued prior to finalizing phase 2.
Groups:
- Omalizumab 150 mg (A): Participants received 150mg omalizumab every 4 weeks during the initial dosing phase (24 weeks). A second dosing period (at 150mg or 300mg) may have been implemented based on protocol-defined assessment criteria.
- Maintained Response (A1): omalizumab 150 mg maintained response group
- Omalizumab 300 mg (B): Participants received 300mg omalizumab every 4 weeks during the initial dosing phase (24 weeks). A second dosing period may have been implemented based on protocol-defined assessment criteria.
- Maintained Response(B1): omalizumab 300 mg Maintained Response group
Arm/Group | Omalizumab 150 mg (A) | Maintained Response (A1) | Retreatment (A2) | Step-up Treatment Group (A3) | Omalizumab 300 mg (B) | Maintained Response(B1) | Retreatment (B2) | Extended Treatment (B3)
Serious Adverse Events (participants affected / at risk) | 2/178 | 0/15 | 0/12 | 2/141 | 6/136 | 2/44 | 2/44 | 1/43
Other Adverse Events (participants affected / at risk) | 119/178 | 9/15 | 10/12 | 94/141 | 109/136 | 32/44 | 37/44 | 37/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab 150 mg (A) (N=178) | Maintained Response (A1) (N=15) | Retreatment (A2) (N=12) | Step-up Treatment Group (A3) (N=141) | Omalizumab 300 mg (B) (N=136) | Maintained Response(B1) (N=44) | Retreatment (B2) (N=44) | Extended Treatment (B3) (N=43)
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Porphyria acute (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.0001% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab 150 mg (A) (N=178) | Maintained Response (A1) (N=15) | Retreatment (A2) (N=12) | Step-up Treatment Group (A3) (N=141) | Omalizumab 300 mg (B) (N=136) | Maintained Response(B1) (N=44) | Retreatment (B2) (N=44) | Extended Treatment (B3) (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Basedow's disease (Endocrine disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye oedema (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia eye (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 5 | 2 | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breath odour (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 1 | 3 | 4 | 1 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 3 | 1 | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Mouth swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 1 | 0 | 8 | 8 | 2 | 1 | 5
Noninfective gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Reflux gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 3 | 0 | 0 | 3 | 2 | 0 | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1 | 1 | 2 | 1 | 0 | 0 | 1
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 2 | 3 | 0 | 2 | 1
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 4 | 3 | 0 | 1
Drug ineffective (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 12 | 1 | 0 | 11 | 6 | 2 | 1 | 3
Granuloma (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 3 | 0 | 0 | 3 | 5 | 0 | 2 | 3
Injection site bruising (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 5 | 2 | 0 | 3 | 2 | 0 | 2 | 0
Pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 1
Polyp (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 2 | 3 | 1 | 1 | 1
Burn infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 3 | 1 | 0 | 2 | 2 | 0 | 2 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 2 | 3 | 1 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 6 | 1 | 2 | 3
Gingivitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Infection parasitic (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 9 | 0 | 0 | 8 | 4 | 3 | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 2 | 2 | 1 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 29 | 3 | 3 | 20 | 24 | 5 | 10 | 8
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 3 | 0 | 0 | 3 | 1 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 4 | 0 | 0 | 4 | 3 | 2 | 1 | 0
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 3 | 1 | 2 | 0
Pulpitis dental (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 3 | 1 | 0 | 2 | 2 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 3 | 0 | 1 | 2 | 5 | 1 | 4 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 10 | 1 | 1 | 8 | 6 | 4 | 1 | 1
Tinea pedis (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 1 | 0 | 1 | 2 | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 2
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 9 | 2 | 2 | 5 | 15 | 4 | 8 | 2
Urinary tract infection (Infections and infestations) | 6 | 1 | 0 | 5 | 6 | 3 | 0 | 3
Vaginal infection (Infections and infestations) | 2 | 0 | 0 | 2 | 2 | 0 | 2 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 5 | 1 | 0 | 4 | 4 | 1 | 3 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 3 | 1 | 2 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 4 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spirometry abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 1 | 0 | 7 | 10 | 4 | 3 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1 | 1 | 5 | 7 | 2 | 1 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 2 | 1 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 3 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 3 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 5 | 2 | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 2 | 5 | 1 | 2 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Oral fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cluster headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 1 | 2 | 6 | 1 | 2 | 3
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 23 | 2 | 2 | 18 | 19 | 5 | 5 | 9
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Migraine (Nervous system disorders) | 2 | 0 | 0 | 2 | 3 | 0 | 1 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 0 | 1 | 3 | 1 | 0 | 0 | 1
Emotional distress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 8 | 0 | 0 | 7 | 3 | 1 | 2 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 2 | 2 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 3 | 4 | 6 | 3 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 1 | 3 | 2 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 6 | 3 | 1 | 0 | 2
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 3 | 0 | 2 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 2 | 2 | 0 | 1 | 1
Chloasma (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 5 | 2 | 2 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 3 | 2 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 4 | 1 | 2 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 4 | 0 | 2 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 3 | 1 | 0 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 9 | 0 | 0 | 8 | 11 | 3 | 3 | 5
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperaemia (Vascular disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 0 | 1 | 1 | 5 | 1 | 2 | 2
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.